CLINICAL TRIAL: NCT04075422
Title: Bezlotoxumab - in "Real Life" - During the First Episode of Clostridium Difficile Infection in Patients With High Risk of Recurrence. BEFORE Study
Brief Title: Bezlotoxumab - in "Real Life" - During the First Episode of Clostridium Difficile Infection in Patients With High Risk of Recurrence.
Acronym: BEFORE
Status: Completed | Type: Observational
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GEIRAS-GIH 0118; SEI-BEZ-2018-01 (Other: AEMPS)
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — bezlotoxumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Prospective cohort: 64 patients treated with Bezlotoxumab
  Interventions: Drug: Bezlotoxumab Injection [Zinplava]
- Retrospective Cohort (Control): All the first episodes diagnosed in each participating sites during the previous year that meet the inclusion criteria

INTERVENTIONS:
Drug: Bezlotoxumab Injection [Zinplava] — Treatment with bezlotoxumad according to the routine clinical practices
  Groups: Prospective cohort

SUMMARY:
The main hypothesis of the study is that Bezlotoxumab is well tolerated and effective in reducing the recurrence of ICD (Clostridium Difficile infection) in patients with a high risk of recurrence in the first episode of ICD.

As a consequence, the number of readmissions and hospital stays, will be reduced in patients treated with Bezlotoxumab.

DETAILED DESCRIPTION:
This is a comparative study of patients with a high risk of recurrence of ICD in the first episode, treated with Bezlotoxumab (together with standard ICD therapy), with patients with first episode of ICD from a paired retrospective cohort (1: 2) using a propensity score.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have granted the IC and who are going to comply with the study visits and procedures according to their life expectations.
* Patient ≥ 18 years of age
* Having a first episode of DCI and presenting an estimated recurrence risk greater than 35%.

Exclusion Criteria:

* Patients <18 years old
* Pregnant or lactating women
* Women of childbearing age who are not willing to use an appropriate contraceptive method (such as oral contraceptives, intrauterine device or contraceptive barrier method along with spermicide or surgical sterilization) during the study.
* Life expectancy less than 6 months
* Impossibility or serious difficulties of clinical follow-up
* Any digestive disease that, at the discretion of the researcher, makes it difficult to assess the response due to impaired bowel habits.
* Immunoglobulin treatment in the last 3 months
* Previous treatment with Bezlotoxumab
* Treatment with an experimental drug in the previous 30 days or participating or planning to participate in any other clinical trial with an experimental drug during the 12-week trial period.
* Anti- ICD treatment forecast for more than 14 days (eg vancomycin in descending pattern) for the current episode.
* Health center staff
* Direct family members of the research team

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective cohort: patient with a high risk of recurrence during the first episode of Clostridium difficile infection.
  Retrospective cohort: all the patients diagnostic of the first episode of clostridium in the previous year and meet the inclusión/exclusión criteria
Sampling Method: Non-Probability Sample
Enrollment: 869 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | Wee 8
  % of patients who, having presented cure of the episode of ICD, develop recurrence of ICD after the treatment of the first episode.
Recurrence rate | Week 24
  % of patients who, having presented cure of the episode of ICD, develop recurrence of ICD after the treatment of the first episode.
Rate of healing of the ICD episode defined as absence of diarrhea within 48 hours after the end of the episode treatment. | 48 hours after the end of the episode treatment
Hospital stays | Throughout the study until 24 weeks after the diagnosis of ICD
  Total days of hospitalization of patients
Percentage of readmissions due to ICD | From the 'Treatment visit' up to week 24 post -treatment visit ( an average of 24 weeks)
Adverse events related with the infusion | 2 hours (1 hour during the infusion and 1 hour post infusion)
  Rate of adverse events. Sampson criteria will be used to define anaphylaxis will be used
Rate of cardiological safety events. | Throughout the study completion, an average of 26 weeks
  Episodes of acute coronary síndrome, arrhythmia, heart failure Will be recorded

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Fundacion de Alcorcón, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Univ. La Paz, Madrid
  - Hospital Univ. Puerta de HIerro, Madrid

IPD SHARING:
Plan to Share IPD: No